CLINICAL TRIAL: NCT04028804
Title: Imaging Cell Proliferation With FLT PET: A Pilot Study in Paediatric Lymphoma Patients With Equivocal FDG PET Findings
Brief Title: FLT PET: A Pilot Study in Lymphoma Patients
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Amer Shammas, Nuclear Medicine Radiologist, The Hospital for Sick Children
Other Study IDs: 1000021766
Record Dates: First submitted 2014-05-12; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Possitron Emission Therapy (PET); FDG PET; FLT PET; Pediatrics
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FDG PET: FDG PET imagaing
  Interventions: Procedure: FDG PET; Procedure: FLT PET
- FLT PET: FLT PET imaging
  Interventions: Procedure: FDG PET; Procedure: FLT PET

INTERVENTIONS:
Procedure: FDG PET — Each patient will receive a single intravenous injection of FDG (5.18 MBq/kg (0.14 mCi/kg)) using a minimum dose of 37 MBq (1 mCi) up to a maximum of 370 MBq (10 mCi) with an accepted 10%-20% variation since dose variation can occur when small concentrated volumes of FDG are being drawn up or radioactive decay has reduced the amount of available.
  Other Names: 2-[fluorine-18]-fluoro-2-deoxy-D-glucose (FDG)
Procedure: FLT PET — The FLT PET scan will be performed 1-5 days after FDG PET in order to ensure consistency between imaging findings. Each patient will receive a single intravenous injection of FLT (5.18 MBq/kg (0.14 mCi/kg)) using a minimum dose of 37 MBq (1 mCi) up to a maximum of 370 MBq (10 mCi) with an accepted 10%-20% variation since dose variation can occur when small concentrated volumes of FLT are being drawn up or radioactive decay has reduced the amount of available.
  Other Names: 3'-deoxy-3'-[fluorine-18]-fluorothymidine (FLT)

SUMMARY:
Background: Residual masses on follow-up surveillance imaging are frequently detected in paediatric patients with Hodgkin's lymphoma and non-Hodgkin's lymphoma. The residual mass may consist of inflammatory, fibrous or necrotic tissue, or it could represent residual tumor. In most cases, positron emission tomography (PET) with 2-[fluorine-18]-fluoro-2-deoxy-D-glucose (FDG) is useful for distinguishing tumor from fibrosis. However, FDG is not tumor-specific, and increased accumulation of the tracer may be seen in a variety of benign entities which can give rise to false-positive or equivocal FDG PET findings. Alternatively, the uptake of 3'-deoxy-3'-[fluorine-18]-fluorothymidine (FLT) reflects cellular proliferation, and may prove to be a reliable method in resolving equivocal FDG PET findings. Indeed, several studies have demonstrated that FLT can be safely administered to children, and in some cases be more useful than FDG PET in differentiating between infection or inflammation and malignancy. This study hypothesizes that FLT PET can be used as an adjunct imaging modality in paediatric lymphoma patients with equivocal interim or post-therapy FDG PET findings, and that this technique can provide additional diagnostic information which will be useful in distinguishing fibrotic or necrotic residual mass lesions from those that may be harbouring malignancy.

DETAILED DESCRIPTION:
This is a prospective pilot study evaluating the clinical use of FLT PET in paediatric patients with Hodgkin's lymphoma (HL) or non-Hodgkin's lymphoma (NHL). The overall objective of this trial is to assess the feasibility of using FLT PET as an adjunct imaging modality to follow-up paediatric lymphoma patients whose interim or post-therapy FDG PET scan is interpreted as being equivocal. The primary outcome measure is to obtain a preliminary estimate of the diagnostic performance (including the sensitivity, specificity and accuracy) of adjunct FLT PET. This pilot study will yield sufficient preliminary data to help justify and design a subsequent larger study of FLT PET in paediatric lymphoma patients.

This study is open only to HL and NHL patients whose interim or post-therapy FDG PET scan is interpreted as being equivocal and in whom it is not possible resolve the exam results using other conventional imaging techniques such as CT or MRI. All FLT PET image findings will be presented to the treating physician(s) responsible for managing the care of any patient enrolled in this trial. Treating physicians will continue to use routine practices to resolve equivocal FDG PET findings.

ELIGIBILITY:
Inclusion Criteria:

* SickKids Hospital patient of any gender or race
* Participants who are able to undergo imaging procedures without general anaesthesia or sedation
* Patient's or the patient's parents'/guardians' written informed consent prior to participation
* Previous FDG PET scan with at least one documented equivocal finding (i.e. SUV ≥ 2.0, but < 3.5) and no other finding(s) that is strongly suggestive of malignancy. The lesion(s) must have a minimum size of 1 cm in diameter by any CIM in order to address the spatial resolution limitations of the PET scanner.

Exclusion Criteria:

* Patients who are pregnant or nursing
* Medically unstable or critically ill
* Lack of informed consent

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of Performing FLT PET Imaging: SUVs values | FLT PET performed within 1-5 days of FDG PET. PET/CT image findings were compared in relation to pathology within 1 month (when tissue sampling was performed), additional cross-sectional imaging, and/or clinical follow-up for at least 3 months.
  To assess the feasibility of performing 3'-deoxy-3'-[fluorine-18]-fluorothymidine positron emission tomography (FLT PET) imaging.
  The investigator's goals were to assess the normal tissue distribution of 18F-FLT and to provide standardized uptake values (SUVs) of lesions demonstrating equivocal uptake on 18F-FDG PET/CT and compare SUVs values of FLT and FDG

SECONDARY OUTCOMES:
Diagnostic Performance | PET/CT image findings were compared in relation to pathology within 1 month (when tissue sampling was performed), additional cross-sectional imaging, and/or clinical follow-up for at least 3 months
  To obtain a preliminary estimate of the diagnostic performance of adjunct 3'-deoxy-3'-[fluorine-18]-fluorothymidine positron emission tomography (FLT PET) in identifying malignant Hodgkin's Lymphoma and Non-Hodgkin's Lymphoma lesions which receive an equivocal diagnosis by 2-[fluorine-18]-fluoro-2-deoxy-D-glucose positron emission tomography (FDG PET). Provide standardized uptake values (SUVs) of lesions demonstrating equivocal uptake on 18F-FDG PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Shammas, Md, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada